CLINICAL TRIAL: NCT00767663
Title: Does Pretreatment With Persantin Reduce Periprocedural Troponin-I Release in Patients Undergoing Elective Single Vessel PCI
Brief Title: Persantin Preceding Elective PCI
Acronym: P3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, G. Rongen, G. Rongen MD PhD, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P3
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Coronary Heart Disease; Percutaneous Transluminal Coronary Angioplasty; Atherosclerosis
MeSH Terms: conditions — Coronary Disease; Atherosclerosis | interventions — Dipyridamole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): dipyridamole
  Interventions: Drug: dipyridamole
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: dipyridamole — dipyridamole slow release 200mg twice daily, minimal 3 days pretreatment
  Other Names: persantin
  Arms: 1
Drug: placebo — placebo twice daily, minimal three days pretreatment
  Arms: 2

SUMMARY:
In this study the investigators will investigate whether a short pretreatment (3-7 days) with dipyridamole 200mg twice daily will protect patients against myocardial injury sustained during an elective dotter operation of the coronary arteries (PCI).

The investigators hypothesize that dipyridamole can reduce myocardial injury sustained during elective PCI.

DETAILED DESCRIPTION:
Rationale:

In elective PCI (percutaneous coronary intervention) up to 40% of the patients show an asymptomatic rise in myonecrosis marker troponin-I. This release of troponin-I has been found to represent irreversible myocardial injury and has been related to an increased risk of restenosis and even long-term mortality. Dipyridamole has been proven to induce protection against ischemia reperfusion injury and to reduce risk of cardiovascular death or event in secondary prevention after TIA or CVA.

Objective:

To test the hypothesis that dipyridamole improves tolerance to ischemia reperfusion injury in patients undergoing elective PCI.

Study design:

Double-blind placebo controlled intervention study

Study population:

Patients undergoing elective PCI

Intervention:

pretreatment with dipyridamole (Persantin Retard) 2dd 200mg or placebo.

Main study parameters:

Periprocedural troponin-I release measured 8 hours after PCI.

Bioequivalence study:

before the start of th clinical trial we will perform a bioequivalent study to test whether our study medication (blinded by recapsuling) equals original dipyridamole capsules. 6 Healthy volunteers in a cross-over randomised design will take original dipyridamole 200 mg SR and recapsuled dipyridamole 200mg SR (prepared by the department of pharmacy of the RUNMC). Plasma dipyridamole concentration will be measured frequently and at baseline and 1 and 3 hours after administration of dipyridamole nucleoside transport inhibitions of erythrocytes will be measured, to assess drug activity.

The clinical trial will only be initialized after conformation of bioequivalence of the study medication to the original dipyridamole.

ELIGIBILITY:
Inclusion Criteria:

* Patients accepted for elective single, native vessel (left anterior descending, right coronary artery or ramus circumflexus (LAD, RCA or RCX)) PCI in the RUNMC
* Troponin-I < 0,20 mmol/L at screening
* Signed Informed consent

Exclusion Criteria:

* unstable angina
* recent myocardial infarction (STEMI or non-STEMI), during two weeks prior to inclusion
* 3-Vessel disease as seen on coronary angiogram
* Stenotic lesion in main stem as seen on coronary angiogram
* CABG in medical history
* asthma (recurrent episodes of dyspnoea and wheezing, or usage of prescribed inhalation medication: i.e. corticosteroids or B2-agonists)
* Treatment with insulin
* Use of prescribed oral anticoagulants (coumarin derivates)
* Use of oral corticosteroids
* Use of sulfonylurea derivates (glibenclamide, tolbutamide, gliclazide, glimepiride)
* Use of heparin or low molecular weight heparin
* Use of metformin
* Use of dipyridamole
* Chronic use of Non Steroid Anti-Inflammatory Drugs (NSAID's)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-10; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Cardiac troponin-I | before and 8 hours after PCI

SECONDARY OUTCOMES:
Effect of pretreatment with dipyridamole 2x200mg on biomarkers reflecting vascular inflammation (hs-CRP, PLA2, PTX3, IL-6, adiponectin, MCP-1, MMP-9) | 3 days treatment minimal
Effect of PCI on biomarkers reflecting vascular inflammation (hs-CRP, PLA2, PTX3, IL-6, adiponectin, MCP-1, MMP-9) | before and 8 hours after PCI

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Rongen, MD PhD, Principal Investigator — RUNMC
Locations (2):
- Netherlands (2):
  - RUNMC, Nijmegen
  - Canisius Wilhelmina Hospital, Nijmegen

REFERENCES:
- [Background] Kleiman NS. Measuring troponin elevation after percutaneous coronary intervention: ready for prime time? J Am Coll Cardiol. 2006 Nov 7;48(9):1771-3. doi: 10.1016/j.jacc.2006.08.008. Epub 2006 Oct 17. No abstract available. PMID 17084248
- [Background] ESPRIT Study Group; Halkes PH, van Gijn J, Kappelle LJ, Koudstaal PJ, Algra A. Aspirin plus dipyridamole versus aspirin alone after cerebral ischaemia of arterial origin (ESPRIT): randomised controlled trial. Lancet. 2006 May 20;367(9523):1665-73. doi: 10.1016/S0140-6736(06)68734-5. PMID 16714187